CLINICAL TRIAL: NCT05074693
Title: Mobile Health to Monitor Risk for COVID-19 and Improve Mental Health During the Pandemic
Brief Title: Mobile Health and COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: University of Oklahoma (Other); Oklahoma State University (Other)
Responsible Party: Principal Investigator, Michael J. Zvolensky, Ph.D., Hugh Roy and Lillie Cranz Cullen Distinguished University Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002802
Record Dates: First submitted 2021-10-02; First posted 2021-10-12 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Anxiety Depression
Keywords: COVID-19; Health Disparities; Mobile Health
MeSH Terms: conditions — COVID-19 | interventions — Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EASE App (Experimental): EASE is a intervention designed to address anxiety and depression symptoms in its users through the use of educational videos, tailored messages, and interoceptive exercises designed to help the user overcome negative feelings of stress.
  Interventions: Other: EASE app
- INSIGHT (Control) APP (Other): The Insight app provides users with educational videos on mindfulness and meditation techniques.
  Interventions: Other: INSIGHT (Control) App

INTERVENTIONS:
Other: EASE app — EASE is a mobile intervention designed to reduce ongoing mental health concerns among BLAI individuals with elevated anxiety and/or depressive symptoms by targeting anxiety sensitivity. The EASE app employs a variety of features to educate its users on how to deal with increased levels of stress, anxiety, and depression, and train users on how to better cope with the negative feelings of stress. The app contains a series of on-demand features, including a coping toolkit, stress management trainings, and a series of educational videos designed to teach participants how to better deal with stress. EASE also utilizes Ecological Momentary Assessments (EMAs) to gather information, and provide personalized messages to users in real time. Finally, EASE is outfitted with COVID-19 related elements, including a symptoms tracker (which participants can use to report symptoms of COVID-19 they may be experiencing), and a collection of COVID-19 related food, housing, and job placement resources.
  Arms: EASE App
Other: INSIGHT (Control) App — A standard of care control intervention was developed using the INSIGHT platform. This app contains a library of educational videos that cover topics such as meditation and mindfulness, as well as general stress reduction techniques. Additionally, participants have access to a "Report Distress" feature that enables them to report moments when they are feeling high levels of stress. Finally, participants will be able to report any COVID-19 related symptoms they experience using a COVID-19 symptom tracker feature. Participants assigned to this condition will received 2 daily EMAs, during which they will be prompted to watch one of the aforementioned educational videos.
  Arms: INSIGHT (Control) APP

SUMMARY:
The proposed research focuses on evaluating the mobile application, Easing Anxiety Sensitivity for Everyone (EASE), to improve overall public health that concerns risks and mental health status during the coronavirus disease of 2019 (COVID-19) pandemic and to minimize the existing health disparities among Black, Hispanic and Latino, and American Indian (BLAI) individuals during this time. EASE provides COVID-19 symptom monitoring, exposure management skills, and psychoeducation on stress and it's impact on infection and disease susceptibility. This study aims to compare the effect of EASE to an empirical measurement of standard-of-care digital intervention and to identify the effective mechanisms in EASE.

DETAILED DESCRIPTION:
The objective of the current trial is to address health disparities in access to behavioral health care during the COVID-19 pandemic among BLAI via an adaptation of our established, initially validated, low-cost, mobile application ('app'). Participants (N = 880; 220 Black, 220 Hispanic and Latino, 220 American Indian, and 220 NLW) will be randomized to either our established clinical grade app: Easing Anxiety Sensitivity for Everyone (EASE; n=440; n=110 from each of the 4 race/ethnic groups), or an active standard-of-care control digital mindfulness/meditation intervention for anxiety and depression (n=440; n=110 from each of the 4 race/ethnic groups). The present study will include a baseline assessment, a 3-month intervention period, a 3-month continued assessment period (with access to intervention materials), and 3- and 6-month post-baseline assessments with a qualitative interview via phone or online platform (e.g., Zoom) at the 6-month follow-up for some participants. Due to the high vulnerability for COVID-19 related medical complications in minority populations, all participants will receive our previously developed COVID-19 monitoring and symptoms intervention component that already is in use (see below for details) for the 6-month study period. In addition, all participants will complete two daily EMAs throughout the study period. For EASE participants, EMAs will guide the just-in-time approach to immediate, personalized behavioral health care. We have had success with participants completing EMAs in our prior work (e.g., approximately 70% of all prompted daily EMAs completed over a 6-month period). Consistent with several of our studies (e.g., Smart-T3 R01, Phoenix, Persist), all assessments will be completed remotely via REDCap and InsightTM app

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Self-identify as Black, Latinx, American Indian, or NLW
* Clinically significant anxiety and/or depressive symptoms as evinced by a score of 8 or higher on the Overall Anxiety Severity and Impairment Scale (OASIS) and/or Overall Depression Severity and Impairment Scale (ODSIS)
* Reside in Texas or Oklahoma
* Willing/able to complete EMAs on study provided or personal smartphone for 6-month study period
* Willing and able to complete the 3- and 6-month follow-up assessments via the app and over the phone (i.e., qualitative interview)
* Score ≥ 4 on the REALM-Short Form indicating > 6th grade English literacy level (needed to complete EMAs)

Exclusion Criteria:

* Not fluent in English
* Lifetime or significant cognitive impairment
* Identifying as a race/ethnicity for which the corresponding study cell has been filled

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 822 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zvolensky, Ph.D., Principal Investigator — University of Houston; Michael Businelle, Ph.D., Principal Investigator — University of Oklahoma Health Sciences
Locations (2):
- United States (2):
  - TSET Health Promotion Research Center, Oklahoma City, Oklahoma
  - RESTORE Laboratory: Research on Emotion, Substance Use Treatment Outcomes, Rehabilitation, and Empowerment, Houston, Texas

REFERENCES:
- [Derived] Rhudy JL, Kell PA, Shadlow JO, Lowe TS, Stephens LD, Zvolensky MJ, Garey L, Kendzor DE, Businelle MS. Assessing racial/ethnic differences in sleep-pain relationships using intensive longitudinal modeling among Native Americans. Sleep. 2026 Jan 13;49(1):zsaf216. doi: 10.1093/sleep/zsaf216. PMID 40709831
- [Derived] Garey L, Zvolensky MJ, Gallagher MW, Vujanovic A, Kendzor DE, Stephens L, Cheney MK, Cole AB, Kezbers K, Matoska CT, Robison J, Montgomery A, Zappi CV, Businelle MS. A Smartphone-Based Intervention for Anxiety and Depression in Racially and Ethnically Diverse Adults (EASE): Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Dec 5;11(12):e40713. doi: 10.2196/40713. PMID 36409958

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EASE App | INSIGHT (Control) APP
Started | 413 | 409
Completed | 413 | 409
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EASE App | INSIGHT (Control) APP | Total
Number analyzed (Participants) | 413 | 409 | 822
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.63 (13.0) | 38.05 (12.5) | 38.34 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 269 | 262 | 531
  Male | 144 | 147 | 291
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 104 | 98 | 202
  Not Hispanic or Latino | 309 | 311 | 620
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The analyzed row differs from the Overall because Hispanic or Latino was our fourth racial and ethnic group examined. In total, we analyzed 4 groups: American Indians, Black or African Americans, White, and Hispanic or Latino.
  Participants
    American Indian or Alaska Native | 103 | 105 | 208
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 103 | 103 | 206
    White | 103 | 103 | 206
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 104 | 98 | 202

OUTCOME MEASURES:

1. Primary Outcome: Everyday Impairment
Description: Changes in reported anxiety and depression related impairment experienced in major life sectors (work performance, household maintenance, social interactions, relationships) as measured by study developed items from Baseline to follow-up assessments. This measure was created by the study team and was 4 items rated from 1 (Strongly disagree) to 5 (Strongly agree). The scale is summed for a total score with ranges from 4 to 25, with higher scores indicating greater everyday impairment.
Time Frame: From Baseline to 6-Months
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | EASE App | INSIGHT (Control) APP
Number analyzed (Participants) | 413 | 409
Scores on a scale
  Everyday Impairment at Baseline | 15.65 (2.84) | 15.47 (2.91)
  Everyday Impairment at 6-month | 12.74 (4.54) | 13.23 (4.40)

2. Primary Outcome: Anxiety
Description: Change from Screener in anxiety on the 5-item Overall Anxiety Severity and Impairment Scale (OASIS) at follow-up appointments. The OASIS is made up of 5 items rated on a scale from 0 to 4. The OASIS is summed for a total score, with a range from 0 to 25, with higher scores indicating higher anxiety severity and impairment.
Time Frame: From Screener to 6-Months
Measure: Mean (95% Confidence Interval); unit: Total Score
Arm/Group | EASE App | INSIGHT (Control) APP
Number analyzed (Participants) | 413 | 409
Total Score
  Anxiety at Baseline | 10.63 [10.30 to 10.95] | 10.84 [10.50 to 11.18]
  Anxiety at 6-months | 7.32 [6.90 to 7.74] | 7.59 [7.15 to 8.02]

3. Primary Outcome: Depression
Description: Change from Screener in depression on the 5-item Overall Depression Severity and Impairment Scale (ODSIS) at subsequent follow-up appointments. The ODSIS is made up of 5 items rated on a scale from 0 to 4. The ODSIS is summed for a total score, with a range from 0 to 25, with higher scores indicating higher depression severity and impairment.
Time Frame: From Screener to 6-Month
Measure: Mean (95% Confidence Interval); unit: Total Score
Arm/Group | EASE App | INSIGHT (Control) APP
Number analyzed (Participants) | 413 | 409
Total Score
  Depression at Baseline | 9.74 [9.34 to 10.15] | 9.82 [9.39 to 10.25]
  Depression at 6-month | 6.45 [5.97 to 6.93] | 6.58 [6.08 to 7.09]

4. Secondary Outcome: Perceived Discrimination
Description: The Everyday Discrimination Scale (EDS) is a six-item scale that assesses perceptions of discrimination or unfair treatment. The EDS will be utilized to explore whether perceived racial discrimination functions as a moderator of treatment effects on the primary outcomes listed as primary outcomes. The EDS is summed for a total score, with a range from 0 to 20. Higher scores indicate greater everyday discrimination.
Time Frame: From Baseline to end of study, up to 6 months.
Reporting Status: Not Posted, anticipated posting 2026-06

5. Secondary Outcome: Racial Bias/Discrimination
Description: The Coronavirus Racial Bias Scale (CRBS) is a brief self-report questionnaire that measures levels of perceived racial bias/discrimination due to the COVID-19 pandemic. The CRBS will be utilized to explore whether perceived racial discrimination due to the COVID-19 pandemic functions as a moderator of the EASE effects. The CRBS will be utilized to explore whether perceived racial discrimination due to the COVID-19 pandemic functions as a moderator of treatment effects on the primary outcomes listed as primary outcomes. The CRBS is a mean score, with higher scores indicating greater coronavirus racial bias.
Time Frame: From Baseline to end of study, up to 6 months.
Reporting Status: Not Posted, anticipated posting 2026-06

6. Secondary Outcome: Perceive Social Support
Description: The Perceived Social Support Questionnaire (F-SozU K-6) is a measure of the perceived social support. The F-SozU K-6 is summed for a total score, with a range from 6 to 24. Higher scores indicate greater degrees of social support. The F-SozU K-6 will be utilized to explore whether social support functions as a moderator of the treatment effects on the primary outcomes listed as primary outcomes.
Time Frame: From Baseline to end of study, up to 6 months.
Reporting Status: Not Posted, anticipated posting 2026-06

7. Secondary Outcome: Subjective Social Status
Description: The MacArthur Scale of Subjective Social Status is a measures of perceived social status. The MSSS will be utilized to explore whether perceived social status functions as a moderator of the treatment effects on the primary outcomes listed as primary outcomes. The MSSS is not score but has a range from 0 to 10.
Time Frame: From Baseline to end of study, up to 6 months.
Reporting Status: Not Posted, anticipated posting 2026-06

8. Secondary Outcome: Anxiety Sensitivity
Description: The Short Scale Anxiety Sensitivity Index (SSASI) will be used to explore whether Intervention effects on study outcomes are mediated by reductions in anxiety sensitivity. The SSASI is a total score with a range from 0 to 20, with higher scores indicating greater anxiety sensitivity.
Time Frame: Baseline to end of study, up to 6 months.
Reporting Status: Not Posted, anticipated posting 2026-06

9. Secondary Outcome: Discrimination Burden
Description: The discrimination burden section of the Jackson Heart Study Discrimination Instrument will be used to measure perceived experience of discrimination. The measure is a total score with ranges from 4 to 12. Higher scores indicate higher difficulty living a productive and full life because of perceived experience of discrimination. This measure will be used to assess whether discrimination burden functions as a moderator of the EASE effects.
Time Frame: From Baseline to end of study, up to 6 months.
Reporting Status: Not Posted, anticipated posting 2026-06

10. Secondary Outcome: Fear of COVID-19
Description: The Fear of COIVD-19 scale will be used to explore whether intervention effects on study primary outcomes are mediated by reductions in fear related to the COVID-19 pandemic. The FCV is summed for a total score with a range from 5 to 25. Higher scores indicate greater fear of COVID-19.
Time Frame: Baseline to end of study, up to 6 months.
Reporting Status: Not Posted, anticipated posting 2026-06

11. Secondary Outcome: Acculturation
Description: The Abbreviated Multidimensional Acculturation Scale (AMAS) assesses an individual's level of acculturation to a host culture. The AMAS is a mean score. For questions that ask participants how strongly they feel apart of U.S. culture, higher scores indicate higher levels of acculturation. For questions that ask about their future of origin, higher score indicate lower levels of acculturation. This measure will be used to assess whether acculturation functions as a moderator of the EASE effects
Time Frame: Baseline
Reporting Status: Not Posted, anticipated posting 2026-06

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | EASE App | INSIGHT (Control) APP
All-Cause Mortality (participants affected / at risk) | 0/413 | 0/409
Serious Adverse Events (participants affected / at risk) | 0/413 | 0/409
Other Adverse Events (participants affected / at risk) | 0/413 | 0/409

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT05074693/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT05074693/ICF_001.pdf